CLINICAL TRIAL: NCT00206388
Title: A Phase I Study of Zoledronic Acid (Zometa) With Cyclophosphamide in Children With Recurrent or Refractory Neuroblastoma and Cortical Bone Involvement (NANT 2004-01)
Brief Title: Zoledronic Acid (ZOMETA) With Cyclophosphamide With Neuroblastoma and Cortical Bone Involvement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: New Approaches to Neuroblastoma Therapy Consortium (Other)
Responsible Party: Principal Investigator, Peter Zage, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16758; ZOMETA; NCT00258414 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: NEUROBLASTOMA
Keywords: NEUROBLASTOMA; RECURRENT; REFRACTORY; CORTICAL; BONE
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Zoledronic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zolendric acid with Cyclophosphamide (Experimental): Zometa will be administered intravenously every 28 days beginning on day 0. Cyclophosphamide will be administered daily without interruption (unless toxicity supervenes) beginning day 0. Each course of therapy will be 28 days. On day 0 of each cycle, cyclophosphamide should be given first, followed by Zometa with a separation between the two drugs of at least one hour. All patients are required to take calcium and Vitamin D supplementation for the duration of study participation.
  Interventions: Drug: Zolendric acid; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Zolendric acid — IV, 2mg/m2/dose on day 0
  Other Names: Zometa
Drug: Cyclophosphamide — fixed dose of 25mg/m2/dose days 0-27
  Other Names: CTX, Cytoxan

SUMMARY:
The purposes of this study are:

1. To find the highest dose of monthly intravenous Zometa that can be given with daily low doses of cyclophosphamide by mouth to children with recurrent or refractory neuroblastoma without causing severe side effects.
2. To find out the side effects seen by giving Zometa and cyclophosphamide on this schedule at different dose levels.
3. To measure blood and urine levels of Zometa during treatment
4. To preliminarily evaluate the antitumor activity of Zometa and concomitant oral cyclophosphamide in children with recurrent and/or refractory neuroblastoma within the confines of a Phase I study.
5. To measure the effects of Zometa on markers of bone breakdown found in urine, blood, and bone marrow
6. To measure the effects of Zometa on the immune system.

DETAILED DESCRIPTION:
Zoledronic Acid (Zometa), a new generation, highly potent bisphosphonate used to treat osteoporosis and hypercalcemia of malignancy, is widely used in adult malignancies with potential for bone metastasis such as breast cancer, multiple myeloma and prostate cancer. Bisphosphonates modulate the bone environment by toxicity to osteoclasts resulting in decreased bone resorption. Zometa is the first bisphosphonate to affect both osteolytic and osteoblastic metastatic lesions. In several large randomized studies in adults with recurrent or advanced malignancies, patients randomized to Zometa had delay in progression of bone metastases and less morbidity (skeletal related events) when compared to either placebo or pamidronate. The toxicity profile of Zometa in adults has been tolerable and includes hypocalcemia, temperature rise, and nausea. The most concerning toxicity is decline in renal function that appears to be related to cumulative dose and the dose rate of administration. In our pre-clinical studies bisphosphonates delayed progression of osteolytic lesions in neuroblastoma tumors xenografted into immunocompromised mice while the combination of Zometa with low dose cyclophosphamide appeared to prolong overall survival. The primary aim of this study is to evaluate the maximum tolerated dose of Zometa combined with low dose oral cyclophosphamide in children with recurrent or refractory neuroblastoma. We will also evaluate the pharmacokinetics of Zometa in children with neuroblastoma and examine the effect of Zometa on markers of bone resorption, cytokines and bone-related growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 30 years of age when enrolled on study.
* A diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* High-risk neuroblastoma with at least ONE of the following: 1. Recurrent/progressive disease. 2. Refractory disease (i.e. less than a partial response to frontline therapy). No biopsy is required for eligibility for study. 3. Persistent disease after at least a partial response to frontline therapy (i.e. patient has had at least a partial response to frontline therapy but still has residual disease by MIBG, CT/MRI, or bone marrow). Patients in this category are REQUIRED to have a biopsy of at least one residual site demonstrating viable neuroblastoma.
* Bone disease demonstrated by uptake on MIBG scan. If the patient's tumor is known to be non-avid for MIBG then the patient must have evidence of either new lesions or progression of prior lesions on bone scan or plain radiographs.
* A Karnofsky or Lansky performance status of greater than or equal to 50%. Patients who are unable to walk because of paralysis or tumor pain, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy of greater than 2 months.
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. 1. Must not have received within 3 weeks of entry onto this study (4 weeks if prior nitrosourea). 2. Patients must not have received radiation for a minimum of four weeks prior to study entry at the site of any lesion that was biopsied to document study eligibility. A minimum of six weeks is required following prior large field radiation therapy (ie: TBI, craniospinal therapy, whole abdomen, total lung, or over 50% marrow space). 3. Patients must not have had an autologous stem cell transplant within 3 months of entry onto this study. Patients status post-allogeneic stem cell transplant are excluded. 4. A minimum of six weeks is required following prior therapeutic doses of MIBG. 5. Must not have received factors that support platelet or white cell number or function within 7 days of study entry. 6 Must not have received bisphosphonate therapy.
* Must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study.
* Organ Function Requirements Adequate Bone Marrow Function: a. ANC greater than or equal to 750 b. Platelet count greater than or equal to 50,000, transfusion independent (defined as no platelet transfusion for one week). NOTE: hematologic criteria must be met by all patients, regardless of neuroblastoma involvement in bone marrow. Adequate Renal Function a. Glomerular Filtration Rate of greater than or equal to 70 ml/min/1.73 m2, OR b. Age-adjusted normal serum creatinine for age Adequate Liver Function a. Total bilirubin less than or equal to 1.5 x normal for age, and b. SGPT (ALT) and SGOT (AST) less than 5 x normal for age.
* Ionized serum calcium greater than or equal to 1.0 mmol/L (Patients are allowed to be on calcium supplements if serum calcium is stable)
* Urinalysis with less than or equal to 1+ heme.
* Reproductive Function: Negative serum beta-HCG in females and use of effective contraception in females and males of child-bearing potential.

Exclusion Criteria:

* Status post-ALLOGENEIC stem cell transplant.
* Received prior bisphosphonate therapy.
* Receiving other investigational agents.
* Have an uncontrolled infection.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Pregnancy or breast feeding.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Toxicity | 28 days, lifetime for delayed toxicities
Maximum tolerated dose (MTD) | 28 days

SECONDARY OUTCOMES:
Anti tumor activity | 1-2 months post treatment
Pharmacokinetics | prior to infusion of first dose and 24h post
Biologic activity | during courses 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zage, MD, Principal Investigator — Baylor College of Medicine
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - USCF School of Medicine, San Francisco, California
  - Lucille Salter Packer Children's Hospital, Stanford, California
  - Indiana University-Riley Children's Hospital, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center, Houston, Texas
  - University of Wisconsin Medical Center, Madison, Wisconsin